CLINICAL TRIAL: NCT05287854
Title: Surgery and Virtual Reality: Interest of Virtual Reality in Oncology for Procedures Under Local Anesthesia in the Operating Room
Acronym: BOREV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ICO-2021-14
Record Dates: First submitted 2022-01-18; First posted 2022-03-18 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Cancer
Keywords: Virtual reality; Pain control; Anxiety control; Local anesthesia; Surgery; Operating room; Analgesia Nociception Index (ANI)
MeSH Terms: conditions — Neoplasms; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local anesthesia + Virtual Reality (Experimental): In addition to local standard anaesthesia, patients benefit from a virtual reality session during the operation using a virtual reality headset
  Interventions: Device: Virtual reality headset
- Local anesthesia alone (No Intervention): Patients benefit only from a local anaesthesia is provided according to the standard procedure

INTERVENTIONS:
Device: Virtual reality headset — Once the patient is on the operating table, the nurse proposes the different possible VR scenarios and installs the RV headset and an audio headset.
  Arms: Local anesthesia + Virtual Reality

SUMMARY:
Virtual Reality (VR) is an interactive and immersive technology that allows you to evolve in a three-dimensional environment created by computer. It appeals to the senses of people by reproducing universes close to reality or imaginary. This process is currently the subject of numerous studies in the field of health because it is a non-invasive tool, a non-pharmacological alternative for the management of pain, anxiety and patient satisfaction.

People with cancer can have a complex care pathway with psychological, anxiety-provoking and potentially painful repercussions. It is for these reasons that offering VR in the operating room for certain procedures under local anesthesia would improve the experience and comfort of care.

BOREV study will assess the interest of VR on pain for procedures under local anesthesia in the operating room in the context of cancer care. The software used, called HypnoVR©, is a medical device, developed specifically for the management of anxiety and pain through hypnosis, sophrology and relaxation techniques.

The main objective of this study is to compare the maximum pain felt with and without RV for different oncological surgical procedures performed under local anesthesia including anesthetic procedures and surgical procedures. The secondary objectives that will support this research are: the evaluation of the level of anxiety, the link with the pain component via the Analgesia Nociception Index (ANI), as well as the satisfaction of the patient and the operator.

According to the results obtained, the VR device could lead to a change in practice in the management of patients and thus be offered on a larger scale within the framework of the management of pain and anxiety

DETAILED DESCRIPTION:
Description of the modalities for recruiting :

During the preoperative consultation, the surgeon or anesthesiologist presents the study to the patient with a cancer requiring a surgery under local anesthesia. He gives the patient the consent form to participate in the study.

Once the consent form has been signed by the patient and the investigator, the investigator prescribes a screening test before surgery.

Patients registration and randomization :

Any patient who has signed an informed consent form (ICF) must be registered in the eCRF in order to be assigned a patient number.

Randomization will be centralized and performed via the eCRF. Patients will be randomly assigned (1:1) at the latest on the day of the surgery.

Experimental group : Local anaesthesia + virtual reality versus Control group : Anesthesia only.

Surgery period :

Regardless of the group, all patients :

* Will receive local anaesthesia according to the standard procedure required for the operation
* Hemodynamic parameters will be measured
* Will be questioned before, immediately after, and at a distance from the surgical procedure on their state of anxiety and immediately after the surgical procedure on the maximum pain felt during the procedure,
* Will be questioned on their satisfaction at the end of surgery.

ANI will be measured before, during and after the operation in patients included at the Saint Herblain site.

A virtual reality headset will be positioned on the patient before the start of the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or more
* Patient eligible for surgery under local anaesthesia in the operating room
* Written informed consent obtained from the patient
* Patient has valid health insurance

Exclusion Criteria:

* Surgical procedure requiring complementary anaesthetic products such as intravenous sedation, nitrous oxide
* Patient requiring an epidural, a paravertebral block
* Patient with known allergy(ies) to local anaesthetics
* Patient with schizophrenia, seizure disorder
* For the investigation site with PhysioDoloris monitor (MDMS): Patient with contraindications to ANI monitoring:

Known heart rhythm disorder (complete arrhythmia by atrial fibrillation) Pacemaker Apnea

* Administration of a sedative premedication in the 6 hours before the surgery
* Visually or hearing impaired patient without a hearing aid
* Patient deprived of liberty or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Comparison, between the "local anesthesia + virtual reality" group and the "local anesthesia alone" group, of the maximum subjective pain induced by the surgical procedure | Immediately after surgery
  Maximum subjective pain is measured by a numerical pain scale of 0 to 10. (0 : no pain ; 10 : maximum pain)

SECONDARY OUTCOMES:
Comparison, between the "local anesthesia + virtual reality" group and the "local anesthesia alone" group, of the objective pain induced by the surgical procedure in patients with Analgesia Nociception Index | in preoperative ; during the surgical procedure ; immediate postoperative
  Pain is evaluated in continuous by to the Analgesia Nociception Index (ANI) measured from the PhysioDoloris monitor (MDMS).
  It is a unitless index between 0 and 100, which describes:
  Pain: 0 ≤ ANI ≤ 40 Discomfort/anxiety: 40 < ANI ≤ 65 Comfort/well-being: 65 < ANI ≤ 100
Comparison, between the "local anesthesia + virtual reality" group and the "local anesthesia alone" group, of hemodynamic constants | in preoperative ; during the surgical procedure ; immediate postoperative
  Heart rate, blood pressure and respiratory rate measured by a multiparametric monitor type M540
Comparison, between the "local anesthesia + virtual reality" group and the "local anesthesia alone" group, of anxiety | in preoperative ; immediate postoperative ; within 30 minutes after the surgery
  Anxiety is measured by a visual analogue scale of 0 to 10. (0 : no anxiety ; 10 : maximum anxiety)
Comparison, between the "local anesthesia + virtual reality" group and the "local anesthesia alone" group, of patient satisfaction | immediate postoperative
  Satisfaction is evaluated by a Lickert scale (Absolutely satisfied / Somewhat satisfied / Neither satisfied nor dissatisfied / Somewhat dissatisfied / Absolutely dissatisfied)
Comparison, between the "local anesthesia + virtual reality" group and the "local anesthesia alone" group, of operator of the surgical procedure | immediate postoperative
  Satisfaction is evaluated by a Lickert scale (Absolutely satisfied / Somewhat satisfied / Neither satisfied nor dissatisfied / Somewhat dissatisfied / Absolutely dissatisfied)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - ICO, Angers
  - ICO, Saint-Herblain